CLINICAL TRIAL: NCT04234880
Title: High-resolution Phosphocreatine and Creatine Mapping of Human Muscle and Brain
Status: Recruiting | Type: Observational
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Jiadi Xu, Associate Professor, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Other Study IDs: IRB00072712
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In this study, we aim to develop and validate a noninvasive approach for quantifying and imaging energy metabolism, without contrast agents, on widely available clinical MRI scanners. Briefly, this technique allows specific and selective imaging of the energy metabolite phosphocreatine (PCr), in vivo and non-invasively. PCr is one of the predominant high-energy phosphates present in brain and muscle and one that is altered by common diseases. Although energy metabolism and PCr play a vital role in cellular homeostasis, there currently are no routine diagnostic tests to noninvasively quantify or map the distribution of PCr with clinically acceptable spatial resolution or/and scan time. Here, we demonstrate that the exchangeable guanidinium protons of millimolar concentration PCr can be exploited to detect it via the water signal in MRI with greatly enhanced sensitivity (molar signal) using chemical exchange saturation transfer (CEST) MRI, and its concentration can be quantified using an artificial neural network (ANN). This new technique, dubbed ANNCEST, allowed us to obtain a high-resolution PCr map on human skeletal muscle within 1.5 min, on a 3T clinical MRI scanner equipped with just the standard MRI setup. To put this in a larger perspective, energy metabolism is critical for cell viability and is altered by many common acquired and inherited diseases. ANNCEST is arguably the first to use widely available MRI scanners to noninvasively image tissue energy metabolism of PCr, and thus would have appeal to a broad readership of scientists and clinicians interested in neurology, muscular dystrophies and myopathies as well as cardiology, to name a few.

ELIGIBILITY:
Inclusion Criteria:

Subject must be at least 18 years of age Subject must be willing and able to undergo verbal and written informed consent Healthy subjects will have no history of cardiovascular or peripheral vascular disease, diabetes, claudication or difficulty walking.

Exclusion Criteria:

1.) Unable to understand the risks, benefits, and alternatives of participation and give meaningful consent, 2.) Contraindications to MRI such (eg implanted metallic objects) 3.) Significant cardiovascular (heart failure, significant coronary artery disease, infiltrative or hypertrophic cardiomyopathy, constrictive pericarditis), pulmonary or musculoskeletal or orthopedic disease that significantly limit exercise capacity 4.) Weight greater than 350 lbs (inability to fit in the MRI), 5.) Cognitive or speech impairments that would limit completion of questionnaires or fatigue reporting. 6) Subjects with rest pain, critical limb ischemia will be excluded for the study. 7) Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the greater Baltimore area. 50 gender matched healthy controls will be recruited.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
High-resolution phosphocreatine and creatine mapping of human skeletal muscle and brain | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- F. M. Kirby Center and Johns Hopkins University Medical School, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No